CLINICAL TRIAL: NCT03624504
Title: China Micra Transcatheter Pacing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: China Micra
Record Dates: First submitted 2018-07-13; First posted 2018-08-10 (Actual); Results first posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Bradycardia
Keywords: Transcatheter Pacing System; Micra Implantable Device; Transfermoral Catheter Delivery System
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Micra Implant Group (Experimental): Subjects with implant attempt with the Micra Transcatheter Pacing System (TPS)
  Interventions: Device: Micra Transcatheter Pacing System (TPS)

INTERVENTIONS:
Device: Micra Transcatheter Pacing System (TPS) — Treatment of subjects eligible for the single chamber ventricular pacemaker per study requirements

SUMMARY:
The China Micra Transcatheter Pacing Study is a prospective, multi-center, single arm human clinical trial utilizing Objective Performance Criterion (OPC) to confirm the safety and efficacy profile of the Micra system for regulatory approval in China.

DETAILED DESCRIPTION:
All study sites will be in China. Subjects successfully implanted with the Micra system in all sites will be followed at implant/pre-discharge, 1-month, 3-months, and 6-months, and at 6-month intervals thereafter (if applicable) through study closure. The overall follow-up period of the study will end when the last enrolled patient has 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have a Class I or II indication for implantation of a single chamber ventricular pacemaker according to ACC/AHA/HRS 2008 guidelines and China guideline.
2. Subjects who are willing to participate in study through consent and willing to undergo study specific required procedures with expectancy of geographically stable for follow up duration.
3. Subjects who are at least 18 years of age.

Exclusion Criteria:

1. Subject has an existing or prior pacemaker, ICD or CRT device implant.
2. Subject has unstable angina pectoris or has had an acute myocardial infarction (AMI) in the 30 days prior to eligibility assessment.
3. Subjects with current implantation of neurostimulator or any other chronically implanted device which uses current in the body. Note that a temporary pacing wire is allowed.
4. Subjects with a mechanical tricuspid valve, implanted vena cava filter, or left ventricular assist device (LVAD).
5. Subjects who are morbidly obese and physician believes telemetry communication of ≤5 inches (12.5 cm) could not be obtained with programmer head.
6. Subjects whose femoral venous anatomy is unable to accommodate a 23 French introducer sheath or implant on the right side of the heart (for example, due to obstructions or severe tortuosity) in the opinion of the implanter.
7. Subjects who are considered as unable to tolerate an urgent sternotomy.
8. Subjects with a known intolerance to Nickel-Titanium (Nitinol) Alloy.
9. Subjects for whom a single dose of 1.0mg dexamethasone acetate may be contraindicated.
10. Subjects with a life expectancy of less than 12-months.
11. Subjects who are currently enrolled or planning to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in concurrent trials is only allowed when document pre-approval is obtained from the Medtronic study manager.
12. Pregnant women or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth regulation method or abstinence.
13. Subjects with exclusion criteria required by local law (age or other).
14. Subjects with medical condition which precludes patient from participation in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu Zhang, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (7):
- China (7):
  - Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Ruijin Hospital Affliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Affliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Micra Implant Group: Subjects with implant attempt with the Micra Transcatheter Pacing System (TPS) Micra Transcatheter Pacing System (TPS): Treatment of subjects eligible for the single chamber ventricular pacemaker per study requirements
Period: Overall Study
Arm/Group | Micra Implant Group
Started | 82
Completed | 81
Not Completed | 1
Not completed — Unsuccessful Implant | 1

BASELINE CHARACTERISTICS:
Arm/Group | Micra Implant Group
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.50 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethinic Chinese | 82
Region of Enrollment [Count of Participants; unit: Participants]
  China | 82
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.0 (3.89)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Complications Free Survival Probability
Description: Freedom rate from Micra implant procedure and/or system related major complications through 6 months post implant
Time Frame: 6 months post implant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Micra Implant Group
Number analyzed (Participants) | 82
percentage of participants | 97.6 [90.6 to 99.4]
Statistical Analysis 1: Comparison: Micra Implant Group; Null hypothesis: Major complication free rate at 6 months post-implant is less than or equal to 83% Alternative hypothesis: Major complication free rate at 6 months post-implant is greater than 83%; Test type: Other — Assume expected performance to be 94%. The Objective Performance Criterion (OPC) is set at 83% (same performance threshold in FDA approved global study). Assumes 0.05 significance level, 2-sided, 80% power and 10% study attrition; p = 0.0021, z test, 1-sided — The threshold for significance was 0.05; Kaplan-Meier survival probability (%) = 97.6, 95% CI 2-sided [90.6 to 99.4] — The major complication free rate (i.e. survival probability) was estimated using the Kaplan-Meier method

2. Secondary Outcome: Pacing Capture Threshold (PCT)
Description: Pacing capture threshold @0.24ms pulse width Capture threshold is defined as the minimum electrical stimulus required to consistently capture the heart outside of the myocardial refractory period.
  Pulse width is the duration of the current flow expressed in milliseconds. The pulse width must be long enough for depolarization to disperse to the surrounding tissue.
Time Frame: Implant, Discharge, Month 1, Month 3, Month 6
Population: 81 subjects with successful implant were eligible at follow up for this data. One subject at Month 1 did not have the PCT completed, so the data is not summarized below.
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Micra Implant Group
Number analyzed (Participants) | 81
Volts
  Implant | 0.52 (0.29)
  Discharge | 0.52 (0.43)
  1 Month: number analyzed (Participants) | 80
  1 Month | 0.50 (0.57)
  3 Months | 0.47 (0.30)
  6 Months | 0.50 (0.32)

3. Secondary Outcome: Impedance
Description: Impedance measured from the Micra device Impedance is the opposition to current flow.
Time Frame: Implant, Discharge, Month 1, Month 3, Month 6
Population: 81 subject with successful implant
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | Micra Implant Group
Number analyzed (Participants) | 81
Ohms
  Implant | 873.83 (228.26)
  Discharge | 781.73 (193.85)
  1 Month | 719.38 (142.27)
  3 Months | 659.01 (130.04)
  6 Months | 632.22 (124.68)

4. Secondary Outcome: Sensing Amplitude
Description: R-wave sensing amplitude measured from the Micra device Sensing is the ability of the pacemaker to "see" when a natural (intrinsic) depolarization is occurring.
Time Frame: Implant, Discharge, Month 1, Month 3, Month 6
Population: 81 subjects with successful implant were eligible at follow up for this data. One subject at Month 1 did not have the R-wave sensing amplitude completed, so the data is not summarized below.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Micra Implant Group
Number analyzed (Participants) | 81
mV
  Implant | 9.41 (3.87)
  Discharge | 11.16 (3.88)
  1 Month: number analyzed (Participants) | 80
  1 Month | 13.53 (3.65)
  3 Months | 13.78 (4.05)
  6 Months | 13.87 (4.18)

5. Secondary Outcome: Adverse Device Effect
Description: Adverse event related to the Micra system or implant procedure
Time Frame: From implant attempt to last subject follow-up, ranging from 0 to 14 months
Population: All enrolled patients with an implant attempt
Measure: Count of Participants; unit: Participants
Arm/Group | Micra Implant Group
Number analyzed (Participants) | 82
Participants
  Anaemia | 1
  Arteriovenous fistula | 1
  Bundle branch block right | 3
  Chest pain | 1
  Deep vein thrombosis | 1
  Device pacing issue | 1
  Dizziness | 1
  Myocardial necrosis marker increased | 1
  Oedema peripheral | 1
  Pyrexia | 1
  Thrombocytopenia | 1
  Troponin increased | 1
  Ventricular extrasystoles | 1

ADVERSE EVENTS:
Time Frame: From implant attempt to last subject follow-up, ranging from 0 to 14 months
Description: Subjects will be assessed for AEs at all scheduled and unscheduled visits. All procedure related, system related, accessory related, underlying condition or disease related, and serious AEs will be collected on the electronic Case Report Forms (eCRFs).
Arm/Group | Micra Implant Group
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 12/82
Other Adverse Events (participants affected / at risk) | 8/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micra Implant Group (N=82)
Angina pectoris (Cardiac disorders) | 1 (2)
Angina unstable (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Hepatic angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 2 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micra Implant Group (N=82)
Upper respiratory tract infection (Infections and infestations) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT03624504/SAP_000.pdf
  • Study Protocol (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT03624504/Prot_001.pdf